CLINICAL TRIAL: NCT06213038
Title: An Open-label, Dose-escalation Study to Evaluate the Safety, Preliminary Efficacy, Immunogenicity and Pharmacokinetic Characteristics of SKG0106 Intraocular Solution After Single Intravitreal Injection in Chinese Patients With Neovascular (Wet) Age-related Macular Degeneration
Brief Title: A Clinical Study Evaluating the Safety and Efficacy of SKG0106 in Patients With Neovascular Age-related Macular Degeneration (nAMD)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Youxin Chen (Other)
Responsible Party: Sponsor-Investigator, Youxin Chen, Professor, Peking Union Medical College Hospital
Organization: Peking Union Medical College Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SKG0106-001
Record Dates: First submitted 2024-01-09; First posted 2024-01-19 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Neovascular Age-related Macular Degeneration
Keywords: AMD; wet AMD; wAMD; nAMD

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dose Level 1 (Experimental): SKG0106 One-Time Intraocular Injection Dose Level 1
  Interventions: Genetic: SKG0106
- Dose Level 2 (Experimental): SKG0106 One-Time Intraocular Injection Dose Level 2
  Interventions: Genetic: SKG0106
- Dose Level 3 (Experimental): SKG0106 One-Time Intraocular Injection Dose Level 3
  Interventions: Genetic: SKG0106

INTERVENTIONS:
Genetic: SKG0106 — SKG0106 is a recombinant adeno-associated virus (AAV) vector-based in vivo gene therapeutic product

SUMMARY:
This is a clinical study to evaluate the safety, preliminary efficacy, immunogenicity of SKG0106 in subjects with nAMD.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary and able to sign a dated ICF prior to any study-related procedures and able to complete the study as required by the protocol;
2. Aged ≥ 50 years at screening;

   Study Eye:
3. Diagnosis of nAMD as determined by the PI;
4. Active CNV lesions secondary to age-related macular degeneration (AMD);
5. Subjects must have been responsive to anti-VEGF therapy as assessed by the PI prior to study treatment

Exclusion Criteria:

1. Any active intraocular or periocular infection or active intraocular inflammation (e.g., infectious conjunctivitis, keratitis, scleritis, endophthalmitis, infectious blepharitis, uveitis) in the study eye at baseline;
2. Retinal pigment epithelial tear in the study eye at screening;
3. Current vitreous hemorrhage in the study eye or history of vitreous hemorrhage within 4 weeks prior to baseline;
4. Any condition that, in the opinion of the investigator, may limit visual acuity improvement in the study eye;
5. History of retinal detachment or active retinal detachment in the study eye;
6. Any prior gene therapy.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2023-05-05 (Actual); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
Characteristics of dose limiting toxicities (DLTs) | 4 weeks
Type, severity, and incidence of ocular and systemic adverse events (AEs) | 48 weeks

SECONDARY OUTCOMES:
Mean change from baseline in best corrected visual acuity (BCVA) at each visit BCVA of the study eye is examined by the Early Treatment of Diabetic Retinopathy Study (ETDRS) testing at screening and baseline. | 24 weeks
Mean change from baseline in central subfield thickness (CST) at each visit Spectral domain optical coherence tomography (SD-OCT) will be performed to measure CST at screening and at each visit (prior to study drug injection, if available). | 24 weeks
Mean change from baseline in patient-reported outcome (VFQ-25) scale score at each visit Both the total scale and subscale scores of the VFQ-25 is ranging from 0 to 100, and higher scores mean a better outcome. | 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Youchen Chen, Principal Investigator — Peking Union Medical College Hospital
Locations (3):
- China (3):
  - Peking Union Medical College Hospital, Beijing
  - Eye & ENT Hospital of Fudan University, Shanghai
  - Xin Hua Hospital Affiliated to Shanghai Jiao Tong University School of MedicineXin Hua Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai

IPD SHARING:
Plan to Share IPD: No